CLINICAL TRIAL: NCT01485042
Title: Phase I Dose Escalation of Pazopanib Plus TH-302 in Advanced Solid Tumors
Brief Title: Dose Escalation Study of Pazopanib Plus TH-302
Acronym: PATH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Hurwitz, MD (Other)
Collaborators: National Comprehensive Cancer Network (Network); GlaxoSmithKline (Industry); Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00031123
Record Dates: First submitted 2011-11-30; First posted 2011-12-05 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Solid Tumors
Keywords: Phase 1; pazopanib; TH-302; advanced solid tumors
MeSH Terms: interventions — pazopanib; TH 302

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation (Experimental): This is a Phase 1 dose escalation with an expanded cohort that will enroll at MTD.
  Interventions: Drug: Pazopanib and TH-302

INTERVENTIONS:
Drug: Pazopanib and TH-302 — Pazopanib 800 mg daily TH-302 IV on Days 1, 8, 15 at MTD Subjects will receive this regimen until disease progression.

SUMMARY:
3 STUDY RATIONALE Based upon the above rationale, the investigators propose a phase I study combining Pazopanib with TH-302 in advanced solid tumors. Pazopanib is FDA approved at a dose of 800mg per day. Using this dose ensures consistency with standard clinical use. It also ensures using the dose most likely to induce maximal hypoxia, which in turn will help ensure maximal local activation of TH-302 (a hypoxia activated prodrug). TH-302 can be given as monotherapy at a weekly dose of 575 mg/m2. When TH-302 is combined with full doses of various chemotherapeutics, the recommended dose of TH-302 has ranged from 240 to 480 mg/m2. Little overlapping toxicity between TH-302 and pazopanib is expected. However to ensure patient safety, the starting dose for the combination will be conservative and use the TH-302 dose found safe with the majority of cytotoxic agents, 340 mg/m2 given days 1,8, 15 on an every 28 day cycle.

Using a standard 3+3 design, the investigators will add increasing doses of TH-302 (340 mg/m2, 480 mg/m2, 575 mg/m2 given weekly, 3 weeks on/1 week off (the standard TH-302 dosing schedule) to the full monotherapy dose of pazopanib (800 mg p.o daily) with expected accrual ranging from 12-18 subjects. Once the recommended phase II dose is identified, the investigators will then enroll an expanded cohort of approximately 12-18 (i.e. total of 30 subjects overall) patients to better define the tolerability of this study drug combination.

4 STUDY OBJECTIVES 4.1 Primary

* To define the maximal tolerated dose (if any) and the recommended phase II doses for the combination of pazopanib plus TH-302 in patients with advanced solid tumors 4.2 Secondary
* To describe any dose limiting and non dose-limiting toxicities of this drug combination

DETAILED DESCRIPTION:
STUDY DESIGN 5.1 Study Description This open-label, non-randomized phase I trial is designed to assess the safety, tolerability and maximum tolerated dose (MTD)/recommended phase II dose (RPTD) of TH-302 plus pazopanib in adult subjects with advanced solid tumors.

Patients will be accrued (enrolled) at Duke University Medical Center. Accrued (enrolled) subjects are defined as subjects who give informed consent. Approximately 50 subjects may be enrolled to ensure the trial obtains approximately 30 evaluable subjects.

Evaluable subjects are defined as those subjects who give informed consent, meet inclusion/exclusion screening criteria, received study drug treatment and completed the first cycle of safety assessments or have dose limiting toxicity that precludes completing the full cycle of assessments.

Please note that the number of accrued subjects exceeds the number of evaluable subjects for the following reasons:

1. Screen failures: Subjects with informed consent that do not meet inclusion/exclusion screening criteria.
2. Treated patients: Subjects with informed consent that meet the inclusion/exclusion criteria and received study drug treatment but did not complete the first cycle of safety assessments for primary study end points (e.g. those subjects who have disease progression or inter-current illness).

There will be two stages to this Phase I study. Stage 1 will be the dose escalation component to determine safety and the recommended phase II dose (RPTD) for TH-302 plus pazopanib combination. Dose escalation will begin with cohort 1 and continue as described in Table 5.1.

Stage 2 will be an expanded cohort which will better describe the tolerability and toxicity profile and (2) to further assess biomarkers related to mechanisms of the study agents. The treatment schedule will be as follows:

Table 5.1 Cohort Doses Cohort # subjects Threshold 302 mg/m2, intravenously Days 1, 8, 15 Pazopanib mg, orally daily

* 1 3-6 240 800 Starting Dose

  1. 3-6 340 800
  2. 3-6 480 800
  3. 3-6 575 800 Expanded Cohort 12-18 RPTD 800

     Subjects will be treated on 28 day cycles after satisfying eligibility and screening criteria.

     Intermediate dosing levels may be explored. Toxicity will be assessed every visit and as clinically indicated. Efficacy will be assessed every 2 cycles and as clinically indicated.

     Dose Escalation and Treatment Schema

     The NCI Common Toxicity Criteria version 4.0 will be used to grade adverse events. The following adverse events will be considered dose limiting toxicity (DLT) if occurring during the first cycle of treatment and deemed to be related to study treatment:
* Hematologic toxicity: Any grade 4 neutropenia, thrombocytopenia or anemia or grade ≥ 3 neutropenia or thrombocytopenia lasting over 7 days
* Any grade 3 thrombocytopenia associated with bleeding
* Neutropenic fever
* Nausea,Vomiting or Diarrhea grade 3 and lasting 4 days despite adequate supportive measures
* Grade ≥ 3 ALT or AST elevation > 7 days
* Other non-hematologic toxicity grade 3 excluding alopecia, anorexia, fatigue, hypertension, isolated lab abnormalities (not clinically significant) and/ rare, idiosyncratic reactions to any of the study drugs. Anorexia, fatigue and hypertension will be considered as DLT only if they reach grade 4 or are considered unmanageable.
* Treatment delay of ≥ 14 days for cycle 2 due to unresolved toxicity
* Any treatment-related death or treatment-related hospitalization

Management and dose modifications associated with adverse events are outlined in Sections 9 and 10.

Dose escalation will proceed in Stage 1 within each cohort according to the following scheme:

Number of Patients with DLT at a Given Dose Level Escalation Decision Rule 0 out of 3 Enter 3 subjects at the next dose level.

1 out of 3 Enter 3 more subjects at this dose level. < 1 out of 6 (a) Proceed to the next dose level OR (b) This will be the recommended MTD/RPTD if at highest dose level. > 2 out of 3-6 Dose escalation will be stopped. Three (3) additional subjects will be entered at the next lowest dose level (if only 3 subjects were treated at this level).

* 3 subjects with advanced solid tumors will be accrued at the starting dose level. If no DLTs are seen, 3 subjects will be enrolled in the next dose level.
* Subjects will be monitored for at least one full cycle before advancement to the next dose level.
* If one of three subjects has DLT at a given dose level, then an additional three subjects will be enrolled at that dose level.
* If 1/6 subjects experiences DLT at a given dose level, then escalation will continue to the next dose level.
* If ≥ 2 out of 3-6 subjects have DLT at any dose level, then that dose level will be considered to have unacceptable toxicity, and the next lower dose level will be expanded to 6 patients. In this case, the next lower dose level will be declared as the MTD provided ≤ 1/6 subjects have DLT (otherwise, dose will be further de-escalated). In cases where the only toxicity seen at this lower dose level is Grade ≤ 2, re-escalation for intermediate dosing will be considered. If there is uncertainty about study drug attribution to DLT then re-escalation to full doses is also permitted.
* If > 33% of subjects has DLT at any dose level, then that dose level will be considered to have unacceptable toxicity. The dose level immediately below the one with unacceptable toxicity will be the recommended phase II dose.
* If no unacceptable toxicity is seen at the highest dose level, then the highest dosing regimen will be considered the MTD or the phase II RPTD.
* Up to 6 subjects will be enrolled at MTD to better define tolerability and safety before proceeding to the expanded cohort.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed malignant solid tumor that is refractory to standard therapies, or for which no standard therapies exist, or for whom pazopanib would be considered a therapeutic option.
* Disease must be measurable by RECIST 1.1 criteria (see Appendix 1).
* Age ≥ 18 years
* Karnofsky Performance status ≥ 80% (see Appendix 2)
* Life expectancy of at least 3 months
* Adequate bone marrow function as shown by:

  * ANC ≥ 1.5 x 109
  * Platelets ≥ 100 x 109/L
  * Hemoglobin ≥ 9 g/dL; Erythropoietin and transfusion support is permitted provided treatments are not required more than every 8 weeks. Hemoglobin must be stable above or equal to 9 g/dL for at least 2 weeks prior to day 1of study drug without blood transfusion to maintain hemoglobin level.
* Adequate liver function as shown by:

  * serum bilirubin ≤ 1.5x ULN
  * PT/PTT/INR ≤ 1.5x ULN
  * ALT and AST ≤ 2.5x ULN
* Adequate renal function: creatinine clearance (estimated) ≥ 50 cc/min by Cockroft-Gault or 24 hour urine (see Appendix 6).
* Baseline MUGA or ECHO must demonstrate LVEF ≥ 50%
* TSH, T3 and T4 within normal limits; Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days from day 1 of study drug; both men and women must be willing to use two methods of contraception, one of them being a barrier method during the study and for 6 months after last study drug administration.
* Signed informed consent

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks from day 1 of study drug (including investigational agents, chemotherapy, radiation therapy, antibody based therapy, etc.)
* Patients who:

  * have had a major surgery or significant traumatic injury within 4 weeks from day 1 of study drug,
  * have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or
  * are anticipated to require major surgery during the course of the study.
* Patients who have exhibited hypersensitivity reactions to pazopanib and/or a structural compound, biological agent, or formulation.
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent with the following exceptions:
* Intermittent steroids (not to exceed 4 mg every day) may be used on an as-needed basis
* Patients on physiologic replacement doses of steroids due to adrenal insufficiency for any reason may remain on these medications.
* Topical, inhaled or intra-articular corticosteroids
* Active brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases. Treated, asymptomatic metastases are permitted provided the patient has been off steroids for at least 1 month prior to day 1 of study drug.
* Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or O2 saturation <90% by pulse oximetry after a 2 minute walk or in the opinion of the investigator any physiological state likely to cause systemic or regional hypoxemia.
* Presence of poorly controlled atrial fibrillation (ventricular heart rate >100 bpm)
* Previous history of CVA, TIA, angina pectoris, acute MI or history of recent re-perfusion procedures (e.g. PTCA), pulmonary embolus or untreated deep vein thrombosis (DVT) within 6 months from day 1 of study drug.

NOTE: Subjects with recent DVT who have been therapeutically anti-coagulated for at least 6 weeks are eligible.

* Congestive heart failure (New York Heart Association (NYHA classification, see Appendix 4 functional classification III-IV).
* Proteinuria at screening demonstrated by urine analysis (UA) > 1+ or 24 hour urine protein ≥ 1 gram/24 hours.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study as so judged by the treating physician. Examples include but are not limited to:

  * Severely impaired lung function (e.g. use of home O2, history of Idiopathic Lung Disease (ILD), any evidence of ILD on scan.
  * Active or uncontrolled severe infections requiring treatment with antibiotics.
  * Liver disease
  * Poorly controlled hypertension [defined as systolic blood pressure (SBP of >140 mmHg or diastolic blood pressure (DBP) of >90 mmHg] NOTE: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Following antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals. At least 24 hours must have elapsed between anti-hypertensive medication initiation or adjustment and BP measurement.
  * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of oral medications (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to day 1 of study drug
* History of hemoptysis within 1 month prior to day 1 of study drug.
* History of abdominal fistula or gastrointestinal perforation at any point within 6 months prior to day 1 of study drug, unless surgically repaired.
* Active peptic ulcer disease inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation or gastrointestinal bleeding.
* Use or need for full dose anticoagulation other than low molecular weight heparin (e.g. Lovenox and no other bleeding risk).
* Invasion or encasement of a major artery. Abutment without invasion or encasement is permitted.
* Serious, non-healing wound, active ulcer, or untreated bone fracture as judged by treating physician.
* Active, bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.
* Known history of HIV or Hepatitis B or C seropositivity.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Two acceptable forms of contraceptives must be continued throughout the trial by either sex. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to day 1 of study drug).
* Concomitant use of CYP3A4 inducers, strong inhibitors or substrates with a narrow therapeutic window.
* Corrected QTc interval > 480 msec. If QTc interval is > 480 msec, then 2 additional ECGs should be obtained over a brief period of time (e.g., within 15-20 minutes) to confirm the abnormality.
* Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose | 12-18 months
  To define the maximal tolerated dose (if any) and the recommended phase II doses for the combination of pazopanib plus TH-302 in patients with advanced solid tumors

SECONDARY OUTCOMES:
Dose limiting or non dose limiting toxicities | 12-18 months
  To describe any dose limiting and non dose-limiting toxicities of this drug combination

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I Hurwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States